CLINICAL TRIAL: NCT05542199
Title: Food Supplement Approach for Prevention of Age-associated Cognitive Decline in Older Adults With Obesity: the Nutrition for Brain and Body Health (BB-Health) Feasibility Trial
Brief Title: Nutrition for Brain and Body Health (BB-Health) Feasibility Trial
Acronym: BB-Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Massachusetts General Hospital (Other); University of Florida (Other); University of New Hampshire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2273
Record Dates: First submitted 2022-08-09; First posted 2022-09-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2023-09

CONDITIONS: Cognition; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: A 2x2 factorial design in which participants are assigned to the multicomponent nutrition supplement or a placebo, and to participation in a behavioral weight loss intervention or to a wait-list control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking occurs after randomization. Participants and investigators and outcome assessors are masked to the assignment to the nutritional supplement vs placebo. Investigators responsible for the weight loss intervention, and outcome assessors, are masked to the assignment to the behavioral weight loss intervention versus the wait-list control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- +MCNS+WL (Active Comparator): This group receives the multicomponent nutrition supplement and the behavioral weight loss intervention.
  Interventions: Other: Multicomponent nutrition supplement (MCNS); Behavioral: Behavioral weight loss program
- -MCNS+WL (Placebo Comparator): This group receives the placebo nutrition supplement and the behavioral weight loss intervention.
  Interventions: Behavioral: Behavioral weight loss program
- +MCNS-WL (Active Comparator): This group receives the multicomponent nutrition supplement and is in the control group for the behavioral weight loss intervention (no behavioral intervention during the trial, but participant is wait-listed to receive one after the trial finishes).
  Interventions: Other: Multicomponent nutrition supplement (MCNS)
- -MCNS-WL (No Intervention): This group receives the placebo nutrition supplement and is in the control group for the behavioral weight loss intervention (no behavioral intervention during the trial, but participant is wait-listed to receive one after the trial finishes)

INTERVENTIONS:
Other: Multicomponent nutrition supplement (MCNS) — Palatable daily nutrition supplement for 12 months containing approximately 300 kcal and a wide range of nutrients and plant constituents with potential to support brain health and cognition.
  Arms: +MCNS+WL; +MCNS-WL
Behavioral: Behavioral weight loss program — Enrollment in behavioral weight loss intervention for 12 months modeled on the Diabetes Prevention Program.
  Arms: +MCNS+WL; -MCNS+WL

SUMMARY:
The goal of the trial is to determine the feasibility of implementing a specific nutrition regimen used alone or in combination with a behavioral weight loss (WL) intervention on cognition and cerebral blood flow in older adults at risk of cognitive decline.

ELIGIBILITY:
Major inclusion criteria:

1. Adult women and men aged 55-85 years.
2. BMI of 27.0-39.9 kg/m2 at screening (higher BMIs not included at this time to facilitate program adherence);
3. Scores of 34 or greater on the Modified Telephone Interview for Cognitive Status (TICS-M) at screening (85). The purpose of this screen is to ensure that participants can give consent and adhere to the study requirements, including the outcomes testing.
4. Willing to be randomized and participate in all study components, including consuming the foods and supplements, participating in the WL intervention or control meetings, being available for outcome assessments, using the provided home Wi-Fi scale and activity monitor daily, and completing questionnaires, as well as providing the login information for scales and activity monitor so investigators can download the data.
5. Satisfactory screening review of health history questionnaire by nursing staff for relevant factors including no evidence of exclusions listed below. This will include verbal confirmation of completing a course of vaccination against COVID-19 (two doses plus one booster prior to screening visit). The reason for this study component is that live group meetings are planned with other participants, and this will reduce participant risk.
6. Has access to computer or smartphone with Wi-Fi and possesses a freezer at home with space for supplement storage.
7. Rates representative food with characteristics of the MCNS and control foods at least 4 on a 5-point scale of liking at screening, and reports that they are willing to consume the food daily.
8. Average energy intake in 3 24-h dietary recalls is within physiological (i.e., plausible) range.

Major exclusion criteria:

1. >25% percentile in most recent data for US adult population intake for reported DHA/EPA in screening questionnaire for rich food sources, which is equivalent to 2 or more servings of fatty fish/month (86, 87).
2. Regularly taking a multivitamin, cacao/cocoa supplement, choline supplement, DHA/EPA supplement, or any supplement advertised for brain health or cognitive function (>1/week). Washout period of 2 months accepted.
3. Does not like, or alternatively reports eating >1 serving per week of >60% chocolate or cocoa.
4. Severe cardiovascular disease including stroke, heart failure, coronary bypass and valve replacement, coronary bypass or any surgical procedures or signs and symptoms of current severe cardiovascular disease.
5. History of neurological brain disease, including stroke, seizure disorders, traumatic brain injury (moderate to severe); including prior diagnosis of a neurodegenerative disease including AD and Parkinson's disease, frontotemporal dementia. Moderate traumatic brain injury is defined by an injury with loss of consciousness.
6. Major psychiatric disorder history (schizophrenia, bipolar affective disorder, intractable depression).
7. Inadequately controlled hypertension at the discretion of study MD or RN
8. Diabetes Type 1 & Type 2 or use of any pharmacological treatment for diabetes or HbA1c >6.5 at screening.
9. Any disorder, unwillingness, or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardize the subject's safety or compliance with the protocol. This includes the lost of smell or taste.
10. History of stomach or bowel resection (other than appendectomy), gastric bypass, or other bariatric weight loss procedure
11. GI diseases, conditions or meds known to influence GI absorption including active peptic ulcer disease or inflammatory bowel disease (such as ulcerative colitis, Crohn's disease), Celiac disease, Cystic Fibrosis, malabsorption disorders, gallbladder disease, acute or chronic pancreatitis or Pancreatic insufficiency
12. Chronic kidney disease or history of kidney stones
13. History of diagnosed eating disorder anorexia, bulimia or binge-eating
14. Active treatment for cancer (except non-melanoma skin cancer) of any type in ≤ 3 year.
15. Thyroid disease or other significant endocrine disorder
16. Uncontrolled hypercholesterolemia.
17. History of acute or chronic pancreatitis or gall bladder disease.
18. Metabolic disorders or conditions that interfere with nutrient absorption (such as Phenylketonuria, Maple Syrup Urine Disease, glucose-galactose malabsorption, ornithine transcarbamylase deficiency or hypophosphatemic rickets.)
19. Dose adjustment to statin or antihypertensive medication within the past 3 months
20. Screening lab results outside the normal parameters that may interfere with study outcomes at the discretion of study MD
21. Inadequate venous access or history of a bilateral mastectomy with nodal dissection
22. Recent history of inflammatory diseases (for example: rheumatoid arthritis, lupus)
23. Active WL, or weight change > 4 kg in past 6 months.
24. Consuming a restrictive diet (e.g. gluten-free, vegan, Paleolithic diet).
25. Self-reported allergy to any ingredient in the provided intervention foods.
26. Self-reported severe allergy to adhesives.
27. Unwilling to use a mobile phone or computer with videoconference software to participate in intervention group meetings. Unwilling to eat on camera.
28. Reports of consumption of > 2 alcoholic drinks per day on average or >14/week (168oz beer/56oz wine/14oz hard liquor.)
29. Reports of consumption of > 2 cups of green or black tea per day on average.
30. Reports of use of recreational and/or illegal drugs.
31. Regular smoking or vaping tobacco or marijuana including the use of edibles within the last 6 months (greater than once a week)
32. Non-English speakers.
33. No social security number (required for stipend payment).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Measure at baseline (pre-randomization), and 3, 6 and 12 months after randomization
  Change in age-sensitive cognitive composite z-score from baseline, based on well-established standardized scores on 5 neuropsychological tests (Controlled Oral; Word Association Test, Digit Symbol Substitution Test; Stroop Interference Test; Trails Making Tests A and B)

SECONDARY OUTCOMES:
Microvascular cerebral blood flow in fasting state | Measure at baseline (pre-randomization), and 3, 6 and 12 months after randomization
  Change in microvascular cerebral blood flow from baseline, measured with diffuse correlation spectroscopy / near infrared spectroscopy during fasting state
Microvascular cerebral blood flow in fed state | Measure at baseline (pre-randomization), and 3, 6 and 12 months after randomization
  Change in microvascular cerebral blood flow from baseline, measured with diffuse correlation spectroscopy / near infrared spectroscopy during fed state
Macrovascular cerebral blood flow velocity in fasting state | Measure at baseline (pre-randomization), and 3, 6 and 12 months after randomization
  Change in macrovascular cerebral blood flow velocity measured with transcranial Doppler ultrasound measured during fasting state
Macrovascular cerebral blood flow velocity in fed state | Measure at baseline (pre-randomization), and 3, 6 and 12 months after randomization
  Change in macrovascular cerebral blood flow velocity measured with transcranial Doppler ultrasound measured during fed state

OTHER OUTCOMES:
Weight loss | Measure at baseline (pre-randomization), and 3, 6 and 12 months after randomization
  Change in body weight from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Susan B. Roberts, Ph.D., Principal Investigator — Jean Mayer USDA Human Nutrition Research Center on Aging
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared consistent with NIH policies.
Time Frame: Within 12 months of publication of the primary paper.